CLINICAL TRIAL: NCT03343067
Title: A Study to Evaluate Safety and Efficacy of Elagolix Alone or Elagolix With Hormonal Add-Back in Subjects With Endometriosis With Associated Moderate to Severe Pain
Brief Title: A Study to Evaluate Safety and Efficacy of Elagolix in Participants With Endometriosis With Associated Moderate to Severe Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early for business reasons, not for safety concerns.
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-383
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-07

CONDITIONS: Endometriosis
Keywords: Endometriosis associated pain; Elagolix; Non-menstrual pelvic pain (NMPP); Dysmenorrhea (DYS)
MeSH Terms: conditions — Endometriosis; Dysmenorrhea | interventions — elagolix; Estradiol; Norethindrone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (Experimental): Day 1 Through Month 3 (Open-Label): Open-Label elagolix 150 mg QD
  Month 4 Through Month 24 (Double-Blind): Efficacy responders to elagolix 150 mg QD at Month 3 and continue treatment through Month 24
  Interventions: Drug: elagolix
- Arm C (Experimental): Day 1 Through Month 3 (Open-Label): Open-Label elagolix 150 mg QD
  Month 4 Through Month 24 (Double-Blind): Incomplete efficacy responders to elagolix 150 mg QD at Month 3 and randomized to elagolix 200 mg BID plus E2/NETA 1/0.5 mg QD treatment group and continue treatment through Month 24.
  Interventions: Drug: elagolix; Drug: estradiol/norethindrone acetate (E2/NETA)
- Arm D (Experimental): Day 1 Through Month 3 (Open-Label): Open-Label elagolix 150 mg QD
  Month 4 Through Month 6 (Double-Blind): Incomplete efficacy responders to elagolix 150 mg QD at Month 3 and randomized to elagolix 150 mg QD treatment group
  Month 7 Through Month 24 (Double-Blind): Incomplete efficacy responders to elagolix 150 mg QD at Month 6 and assigned to elagolix 200 mg BID plus E2/NETA 1/0.5 mg QD treatment group and continue treatment through Month 24.
  Interventions: Drug: elagolix; Drug: estradiol/norethindrone acetate (E2/NETA)
- Arm B (Experimental): Day 1 Through Month 3 (Open-Label): Open-Label elagolix 150 mg QD
  Month 4 Through Month 6 (Double-Blind): Incomplete efficacy responders to elagolix 150 mg QD at Month 3 and randomized to elagolix 150 mg QD treatment group
  Month 7 Through Month 24 (Double-Blind): Efficacy responders to elagolix 150 mg QD at Month 6 and continue treatment through Month 24.
  Interventions: Drug: elagolix

INTERVENTIONS:
Drug: elagolix — Tablets
Drug: estradiol/norethindrone acetate (E2/NETA) — Capsules
  Arms: Arm C; Arm D

SUMMARY:
This is a Phase 3, dose-escalation study designed to evaluate the safety and efficacy of both elagolix alone and elagolix plus estradiol/norethindrone acetate (E2/NETA) over 24 months in the management of endometriosis with associated moderate to severe pain in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a premenopausal female 18 to 49 years of age (inclusive) at the time of Screening.
* Participant has a documented surgical diagnosis (e.g., laparoscopy or laparotomy) of endometriosis established by visualization or histology within 10 years prior to entry into Washout or Screening,
* Participant must agree to use only those rescue analgesics permitted by the protocol during the Screening and Treatment Periods for her endometriosis-associated pain.
* Participant must have the following documented in the e-Diary during the last 35 days prior to Study Day 1:

  1. At least 2 days of "moderate" or "severe" DYS, AND either,
  2. At least 2 days of "moderate" or "severe" NMPP and an average NMPP score of at least 1.0, OR
  3. At least 4 days of "moderate" or "severe" NMPP and an average NMPP score of at least 0.5.

Exclusion Criteria:

* Participant has chronic pelvic pain that is not caused by endometriosis that requires chronic analgesic therapy, which would interfere with the assessment of endometriosis-associated pain.
* Participant is using any systemic corticosteroids for over 14 days within 3 months prior to Screening or is likely to require treatment with systemic corticosteroids during the course of the study. Over-the-counter and prescription topical, inhaled or intranasal corticosteroids are allowed.
* Participant has a history of major depression or post-traumatic stress disorder (PTSD) within 2 years prior to screening or other major psychiatric disorder at any time
* Participant has a history of suicide attempts or answered "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening or prior to study drug dosing on Day 1.
* Participant has any condition that would interfere with obtaining adequate dual energy x-ray absorptiometry (DXA) measurements
* Screening DXA results of the lumbar spine (L1 - L4), femoral neck or total hip bone mineral density (BMD) corresponding to less than 2 or more standard deviations below normal (Z-score < -2.0 for participants < 40 years of age, T-score for participants >= 40 years of age).
* Participant has either

  1. a newly diagnosed, clinically significant medical condition that requires therapeutic intervention (e.g., new onset hypertension) that has not been stabilized 30 days prior to enrollment on Day 1 OR
  2. a clinically significant medical condition that is anticipated to required intervention during the course of study participation (e.g., anticipated major elective surgery) OR
  3. an unstable medical condition that makes the participant an unsuitable candidate for the study in the opinion of the Investigator
* Participant has any conditions contraindicated with use of E2/NETA

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (37):
- United States (37):
  - Pinnacle Research Group /ID# 202016, Anniston, Alabama
  - Noble Clinical Research /ID# 170628, Tucson, Arizona
  - Lynn Institute of the Ozarks /ID# 165052, Little Rock, Arkansas
  - SC Clinical Research /ID# 165049, Garden Grove, California
  - Marvel Clinical Research /ID# 169633, Huntington Beach, California
  - Health care Affiliates Medical Group /ID# 165048, Santa Ana, California
  - Western States Clinical Res /ID# 169809, Wheat Ridge, Colorado
  - Nova Clinical Research, LLC /ID# 202227, Bradenton, Florida
  - Midland Florida Clinical Research Center /ID# 201327, DeLand, Florida
  - Southeastern Integrated Med /ID# 203109, Gainesville, Florida
  - Care Partners Clinical Researc /ID# 168395, Jacksonville, Florida
  - LCC Medical Research Institute /ID# 168888, Miami, Florida
  - A Premier Clinical Research of Florida, LLC /ID# 201887, Orange City, Florida
  - GCP Clinical Research, LLC /ID# 169774, Tampa, Florida
  - Triple O Research Institute /ID# 201128, West Palm Beach, Florida
  - Bingham Memorial Hospital /ID# 170110, Blackfoot, Idaho
  - Leavitt Womens Healthcare /ID# 169495, Idaho Falls, Idaho
  - Quad Clinical Research, LLC /ID# 168294, Chicago, Illinois
  - Quad Clinical Research, LLC /ID# 170629, Chicago, Illinois
  - Women's Health Care, PC /ID# 165033, Newburgh, Indiana
  - Delricht Research /ID# 200219, New Orleans, Louisiana
  - Quad Clinical Research, LLC /ID# 200180, St Louis, Missouri
  - Montana Health Research Inst /ID# 170624, Billings, Montana
  - Excel Clinical Research /ID# 170620, Las Vegas, Nevada
  - Northwell health system /ID# 200162, Manhasset, New York
  - Radiant Research, Inc /ID# 200045, Akron, Ohio
  - Central Ohio Clinical Research /ID# 170750, Columbus, Ohio
  - Optimed Research /ID# 167642, Columbus, Ohio
  - VitaLink Research /ID# 168401, Greenville, South Carolina
  - VitaLink Research /ID# 170625, Greenville, South Carolina
  - Fusion Clinical Research of Spartanburg /ID# 200010, Spartanburg, South Carolina
  - Centex Studies, Inc /ID# 169897, Houston, Texas
  - America's Adv. Wellness Center /ID# 170005, Houston, Texas
  - ClinRx Research, LLC /ID# 201189, Plano, Texas
  - Progressive Clinical Research /ID# 205565, San Antonio, Texas
  - Eastern Virginia Med School /ID# 165016, Norfolk, Virginia
  - Seattle Reproductive Medicine /ID# 171079, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated early for business reasons, not for safety concerns. There are no subject data past Treatment Month 6.
Groups:
- Group A: Day 1 through Month 3 (open-label): elagolix 150 mg QD
  Participants discontinued prematurely during the open-label period.
- Group B: Day 1 Through Month 3 (Open-Label): Open-Label elagolix 150 mg QD
  Month 4 Through Month 6 (Double-Blind): Efficacy responders to elagolix 150 mg QD Month 3 continued on elagolix 150 mg QD
  The efficacy responder status of each participant was determined based on the responses to the Daily Diary endometriosis-associated pain score via a Numeric Rating Scale (NRS) in the electronic diary. Efficacy responder: ≥ 30% decrease (improvement) from Baseline based on the average of the Daily Diary for endometriosis-associated pain score via NRS over a 35 day window.
- Group C: Day 1 Through Month 3 (Open-Label): Open-Label elagolix 150 mg QD
  Month 4 Through Month 6 (Double-Blind): Incomplete efficacy responders to elagolix 150 mg QD at Month 3 and randomized to elagolix 200 mg BID plus E2/NETA 1/0.5 mg QD treatment group
  The efficacy responder status of each participant was determined based on the responses to the Daily Diary endometriosis-associated pain score via NRS in the electronic diary. Incomplete efficacy responder: < 30% decrease (improvement) from Baseline based on the average of the Daily Diary for endometriosis-associated pain score via NRS over a 35 day window
Period: Open Label Period: Day 1 to Month 3
Arm/Group | Group A | Group B | Group C
Started | 7 | 3 | 1
Completed | 0 | 3 | 1
Not Completed | 7 | 0 | 0
Period: Double Blind Period: Month 3 to Month 6
Arm/Group | Group A | Group B | Group C
Started | 0 | 3 | 1
Completed | 0 | 0 | 0
Not Completed | 0 | 3 | 1
Not completed — Study Terminated by Sponsor | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 7 | 3 | 1 | 11
Age, Customized [Count of Participants; unit: Participants]
  20 to < 25 years | 1 | 1 | 0 | 2
  25 to < 30 years | 0 | 1 | 0 | 1
  30 to < 35 years | 1 | 0 | 1 | 2
  35 to < 40 years | 1 | 0 | 0 | 1
  40 to < 45 years | 3 | 1 | 0 | 4
  45 to < 50 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 1 | 11
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 6 | 2 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 5 | 1 | 0 | 6
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Dysmenorrhea (DYS) Pain Scale [Mean (Standard Deviation); unit: score on a scale] — The DYS pain scale score ranged from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe), recorded in a daily eDiary. A minimum of 45 days of daily e-Diary entries were required to be completed during the Screening Period.
  score on a scale | 0.641 (0.1689) | 0.429 (0.1030) | 0.600 (NA) — 1 participant analyzed | 0.579 (0.1696)
Non-Menstrual Pelvic Pain (NMPP) Pain Scale [Mean (Standard Deviation); unit: score on a scale] — The NMPP pain scale score ranged from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe), recorded in a daily eDiary. A minimum of 45 days of daily e-Diary entries were required to be completed during the Screening Period.
  score on a scale | 1.053 (0.4534) | 0.914 (0.4721) | 2.400 (NA) — 1 participant analyzed | 1.138 (0.5893)
Dyspareunia Pain Scale [Mean (Standard Deviation); unit: score on a scale] — The dyspareunia pain scale score ranged from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe), recorded in a daily eDiary. A minimum of 45 days of daily e-Diary entries were required to be completed during the Screening Period. Population: 1 subject did not complete assessment
  score on a scale
    number analyzed (Participants) | 7 | 2 | 1 | 10
    (all) | 0.539 (0.9064) | 0.043 (0.0202) | 3.000 (NA) — 1 participant analyzed | 0.686 (1.1187)
Daily Diary Endometriosis-Associated Pain Score Via Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: score on a scale] — The NRS for overall endometriosis-associated pain ranges from 0 (none) to 10 (worst pain ever), recorded in a daily eDiary. A minimum of 45 days of daily e-Diary entries were required to be completed during the Screening Period.
  score on a scale | 5.176 (1.9302) | 3.638 (1.5692) | 7.371 (NA) — 1 participant analyzed | 4.956 (1.9663)
Rescue Analgesic Use Across Both Classes of Rescue Analgesics (NSAIDs/Opioids) [Mean (Standard Deviation); unit: pills/day] — Based on average pill counts and assessed using the daily e-Diary. Participants were allowed to take protocol-specified analgesic rescue medication for endometriosis-associated pain and recorded use daily in the e-Diary. A minimum of 45 days of daily e-Diary entries were required to be completed during the Screening Period. Permitted non-steroidal anti-inflammatory drugs (NSAIDs) included naproxen, ibuprofen, diclofenac, and celecoxib. Permitted opioids included hydrocodone + acetaminophen and codeine phosphate + acetaminophen.
  pills/day
    NSAID | 2.388 (2.7765) | 0.581 (0.9330) | 0.743 (NA) — 1 participant analyzed | 1.745 (2.3655)
    Opioid | 0.241 (0.3750) | 0.057 (0.0990) | 0.571 (NA) — 1 participant analyzed | 0.221 (0.3270)
    NSAID + Opioid | 2.629 (2.6903) | 0.638 (0.8918) | 1.314 (NA) — 1 participant analyzed | 1.966 (2.3196)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responders at Month 6 Based on DYS Pain Scale
Description: Proportion of responders at Month 6 based upon the scale for DYS pain scale (ranging from 0 [none] to 3 [severe]) using the daily e-Diary, as well as no increased analgesic rescue use for endometriosis-associated pain.
Time Frame: Month 6
Population: Analysis was intended to be based on a receiver operating characteristic (ROC) threshold, which could not be calculated, since only 1 participant had a Month 6 assessment for this endpoint at the time of study termination.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Proportion of Responders at Month 6 Based on NMPP Pain Scale
Description: Proportion of responders at Month 6 based upon the scale for NMPP pain scale (ranging from 0 [none] to 3 [severe]) using the daily e-Diary, as well as no increased analgesic rescue use for endometriosis-associated pain.
Time Frame: Month 6
Population: Analysis was intended to be based on ROC threshold, which could not be calculated, since only 1 participant had a Month 6 assessment for this endpoint at the time of study termination.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in DYS at Month 6
Description: The DYS pain scale score ranged from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe), recorded in a daily eDiary and averaged monthly based on a 35-day window. A negative change from baseline indicates improvement.
Time Frame: Month 0 (baseline), Month 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 1 | 0
score on a scale |  | -0.23 (NA) — 1 participant analyzed |

4. Secondary Outcome: Change From Baseline in NMPP at Month 6
Description: The NMPP pain scale score ranged from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe), recorded in a daily eDiary and averaged monthly based on a 35-day window. A negative change from baseline indicates improvement.
Time Frame: Month 0 (baseline), Month 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 2 | 0
score on a scale |  | -0.13 (0.061) |

5. Secondary Outcome: Change From Baseline in Dyspareunia at Month 6
Description: The dyspareunia pain scale score ranged from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe), recorded in a daily eDiary and averaged monthly based on a 35-day window. A negative change from baseline indicates improvement.
Time Frame: Month 0 (baseline), Month 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 1 | 0
score on a scale |  | 0.29 (NA) — 1 participant analyzed |

6. Secondary Outcome: Change From Baseline in Daily Diary Endometriosis-Associated Pain Score Via Numeric Rating Scale (NRS) at Month 6
Description: The NRS for overall endometriosis-associated pain ranges from 0 (none) to 10 (worst pain ever), recorded in a daily eDiary and averaged monthly based on a 35-day window. A negative change from baseline indicates improvement.
Time Frame: Month 0 (baseline), Month 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 2 | 0
score on a scale |  | -1.36 (0.020) |

7. Secondary Outcome: Change From Baseline in Rescue Analgesic Use Across Both Classes of Rescue Analgesics (NSAIDs/Opioids) at Month 6
Description: Based on average pill counts and assessed using the daily e-Diary. Permitted non-steroidal anti-inflammatory drugs (NSAIDs) included naproxen, ibuprofen, diclofenac, and celecoxib. Permitted opioids included hydrocodone + acetaminophen and codeine phosphate + acetaminophen.
Time Frame: Month 0 (baseline), Month 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: pills/day
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 2 | 0
pills/day
  NSAID: Change at Month 6 |  | 0.63 (0.606) |
  Opioid: Change at Month 6 |  | 0.09 (0.121) |
  NSAID + Opioid: Change at Month 6 |  | 0.71 (0.485) |

8. Secondary Outcome: Percentage of Participants With 30% or More Reduction From Baseline Based on the 35 Day Mean of the Daily Diary Endometriosis-Associated Pain Score Via NRS at Month 6
Description: The NRS for overall endometriosis-associated pain ranges from 0 (none) to 10 (worst pain ever), recorded in a daily eDiary and averaged monthly based on a 35-day window.
Time Frame: Month 6
Population: Participants with both baseline and post-baseline values for Daily Diary Endometriosis-Associated Pain Score via NRS.
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 2 | 0
percentage of participants |  | 50.0 |

9. Secondary Outcome: Proportion of Responders Over Time
Description: As assessed by change and percent change from baseline in average pain score and rescue analgesic use monthly for DYS, NMPP, dyspareunia, and Daily Diary endometriosis-associated pain score via NRS, respectively.
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Analysis was intended to be based on ROC threshold, which could not be calculated for this endpoint due to low enrollment at the time of study termination.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Proportion of Responders Over Time (Not Taking Into Consideration of Analgesic Use)
Description: as for outcome 9
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: as for outcome 9
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline Over Time in Monthly Average DYS Pain Score
Description: The DYS pain scale score ranged from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe), recorded in a daily eDiary and averaged monthly based on a 35-day window. A negative change from baseline indicates improvement.
  The analysis was based on a 28-day window. If a participant prematurely discontinued during the open-label period, based on the analysis window, some data might fall into Month 4 analysis.
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6 | 2 | 0
score on a scale
  Change at Month 1: number analyzed (Participants) | 6 | 1 | 0
  Change at Month 1 | 0.05 (0.655) | -0.04 (NA) — 1 participant analyzed |
  Change at Month 2: number analyzed (Participants) | 4 | 1 | 0
  Change at Month 2 | -0.18 (0.124) | -0.26 (NA) — 1 participant analyzed |
  Change at Month 3: number analyzed (Participants) | 2 | 1 | 0
  Change at Month 3 | -0.50 (0.263) | -0.34 (NA) — 1 participant analyzed |
  Change at Month 4: number analyzed (Participants) | 1 | 1 | 0
  Change at Month 4 | -0.69 (NA) — 1 participant analyzed | -0.06 (NA) — 1 participant analyzed |
  Change at Month 5: number analyzed (Participants) | 0 | 2 | 0
  Change at Month 5 |  | -0.16 (0.141) |
  Change at Month 6: number analyzed (Participants) | 0 | 1 | 0
  Change at Month 6 |  | -0.23 (NA) — 1 participant analyzed |

12. Secondary Outcome: Change From Baseline Over Time in Monthly Average NMPP Pain Score
Description: as for outcome 4
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6 | 3 | 1
score on a scale
  Change at Month 1 | -0.13 (0.252) | -0.07 (0.508) | 0.39 (NA) — 1 participant analyzed
  Change at Month 2: number analyzed (Participants) | 5 | 3 | 1
  Change at Month 2 | -0.48 (0.394) | -0.30 (0.167) | 0.29 (NA) — 1 participant analyzed
  Change at Month 3: number analyzed (Participants) | 2 | 3 | 1
  Change at Month 3 | -0.70 (0.828) | -0.30 (0.092) | 0.54 (NA) — 1 participant analyzed
  Change at Month 4: number analyzed (Participants) | 1 | 3 | 1
  Change at Month 4 | -1.34 (NA) — 1 participant analyzed | -0.34 (0.029) | 0.46 (NA) — 1 participant analyzed
  Change at Month 5: number analyzed (Participants) | 0 | 3 | 0
  Change at Month 5 |  | -0.27 (0.256) |
  Change at Month 6: number analyzed (Participants) | 0 | 2 | 0
  Change at Month 6 |  | -0.13 (0.061) |

13. Secondary Outcome: Change From Baseline Over Time in Monthly Average Dyspareunia Pain Score
Description: as for outcome 5
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 4 | 2 | 1
score on a scale
  Change at Month 1 | -0.50 (0.741) | 0.30 (NA) — 1 participant analyzed | -0.29 (NA) — 1 participant analyzed
  Change at Month 2: number analyzed (Participants) | 2 | 1 | 1
  Change at Month 2 | -1.44 (1.071) | 0.06 (NA) — 1 participant analyzed | -0.37 (NA) — 1 participant analyzed
  Change at Month 3: number analyzed (Participants) | 1 | 2 | 1
  Change at Month 3 | -2.20 (NA) — 1 participant analyzed | 0.07 (0.101) | -0.03 (NA) — 1 participant analyzed
  Change at Month 4: number analyzed (Participants) | 1 | 2 | 1
  Change at Month 4 | -2.23 (NA) — 1 participant analyzed | 0.09 (0.040) | -0.03 (NA) — 1 participant analyzed
  Change at Month 5: number analyzed (Participants) | 0 | 2 | 0
  Change at Month 5 |  | 0.09 (0.081) |
  Change at Month 6: number analyzed (Participants) | 0 | 1 | 0
  Change at Month 6 |  | 0.29 (NA) — 1 participant analyzed |

14. Secondary Outcome: Change From Baseline Over Time in Monthly Average Daily Diary Endometriosis-Associated Pain Score Via NRS
Description: as for outcome 6
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Change at Month 1 | -0.86 (1.975) | -0.89 (1.159) | -0.84 (NA) — 1 participant analyzed
  Change at Month 2: number analyzed (Participants) | 5 | 3 | 1
  Change at Month 2 | -2.40 (2.106) | -2.02 (0.758) | -1.40 (NA) — 1 participant analyzed
  Change at Month 3: number analyzed (Participants) | 2 | 3 | 1
  Change at Month 3 | -3.70 (3.616) | -1.81 (0.430) | -1.34 (NA) — 1 participant analyzed
  Change at Month 4: number analyzed (Participants) | 1 | 3 | 1
  Change at Month 4 | -6.43 (NA) — 1 participant analyzed | -1.43 (1.078) | -1.06 (NA) — 1 participant analyzed
  Change at Month 5: number analyzed (Participants) | 0 | 3 | 0
  Change at Month 5 |  | -1.40 (0.961) |
  Change at Month 6: number analyzed (Participants) | 0 | 2 | 0
  Change at Month 6 |  | -1.36 (0.020) |

15. Secondary Outcome: Percent Change From Baseline to Each Month During the Treatment Period for DYS
Description: as for outcome 3
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: percent change of units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6 | 2 | 0
percent change of units on a scale
  Percent Change at Month 1: number analyzed (Participants) | 6 | 1 | 0
  Percent Change at Month 1 | 1.67 (109.961) | -7.89 (NA) — 1 participant analyzed |
  Percent Change at Month 2: number analyzed (Participants) | 4 | 1 | 0
  Percent Change at Month 2 | -27.45 (17.119) | -75.00 (NA) — 1 participant analyzed |
  Percent Change at Month 3: number analyzed (Participants) | 2 | 1 | 0
  Percent Change at Month 3 | -62.92 (24.159) | -85.71 (NA) — 1 participant analyzed |
  Percent Change at Month 4: number analyzed (Participants) | 1 | 1 | 0
  Percent Change at Month 4 | -80.00 (NA) — 1 participant analyzed | -16.67 (NA) — 1 participant analyzed |
  Percent Change at Month 5: number analyzed (Participants) | 0 | 2 | 0
  Percent Change at Month 5 |  | -40.48 (33.672) |
  Percent Change at Month 6: number analyzed (Participants) | 0 | 1 | 0
  Percent Change at Month 6 |  | -57.14 (NA) — 1 participant analyzed |

16. Secondary Outcome: Percent Change From Baseline to Each Month During the Treatment Period for NMPP
Description: as for outcome 4
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: percentage change of units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6 | 3 | 1
percentage change of units on a scale
  Percent Change at Month 1 | -11.81 (26.677) | 4.22 (53.238) | 16.07 (NA) — 1 participant analyzed
  Percent Change at Month 2: number analyzed (Participants) | 5 | 3 | 1
  Percent Change at Month 2 | -37.53 (31.150) | -34.21 (18.044) | 11.90 (NA) — 1 participant analyzed
  Percent Change at Month 3: number analyzed (Participants) | 2 | 3 | 1
  Percent Change at Month 3 | -38.26 (42.319) | -38.03 (20.343) | 22.62 (NA) — 1 participant analyzed
  Percent Change at Month 4: number analyzed (Participants) | 1 | 3 | 1
  Percent Change at Month 4 | -71.21 (NA) — 1 participant analyzed | -44.49 (20.725) | 19.05 (NA) — 1 participant analyzed
  Percent Change at Month 5: number analyzed (Participants) | 0 | 3 | 0
  Percent Change at Month 5 |  | -28.40 (33.641) |
  Percent Change at Month 6: number analyzed (Participants) | 0 | 2 | 0
  Percent Change at Month 6 |  | -17.23 (16.044) |

17. Secondary Outcome: Percent Change From Baseline to Each Month During the Treatment Period for Dyspareunia
Description: as for outcome 5
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: percentage change of units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
percentage change of units on a scale
  Percent Change at Month 1 | 0.14 (18.180) | -15.27 (26.791) | -9.52 (NA) — 1 participant analyzed
  Percent Change at Month 2: number analyzed (Participants) | 5 | 3 | 1
  Percent Change at Month 2 | 6.60 (15.719) | -15.26 (21.840) | -12.38 (NA) — 1 participant analyzed
  Percent Change at Month 3: number analyzed (Participants) | 2 | 3 | 1
  Percent Change at Month 3 | 60.88 (65.632) | -21.63 (24.719) | -0.95 (NA) — 1 participant analyzed
  Percent Change at Month 4: number analyzed (Participants) | 1 | 3 | 1
  Percent Change at Month 4 | 106.25 (NA) — 1 participant analyzed | -12.67 (20.433) | -0.95 (NA) — 1 participant analyzed
  Percent Change at Month 5: number analyzed (Participants) | 0 | 3 | 0
  Percent Change at Month 5 |  | -14.86 (16.002) |
  Percent Change at Month 6: number analyzed (Participants) | 0 | 2 | 0
  Percent Change at Month 6 |  | -18.08 (25.571) |

18. Secondary Outcome: Percent Change From Baseline to Each Month During the Treatment Period for Daily Diary Endometriosis-Associated Pain Score Via NRS
Description: as for outcome 6
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: percentage change of score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
percentage change of score on a scale
  Percent Change at Month 1 | -14.10 (37.146) | -19.61 (35.468) | -11.34 (NA) — 1 participant analyzed
  Percent Change at Month 2: number analyzed (Participants) | 5 | 3 | 1
  Percent Change at Month 2 | -37.82 (18.066) | -56.25 (4.507) | -18.99 (NA) — 1 participant analyzed
  Percent Change at Month 3: number analyzed (Participants) | 2 | 3 | 1
  Percent Change at Month 3 | -43.98 (35.509) | -53.05 (13.803) | -18.22 (NA) — 1 participant analyzed
  Percent Change at Month 4: number analyzed (Participants) | 1 | 3 | 1
  Percent Change at Month 4 | -70.98 (NA) — 1 participant analyzed | -38.00 (31.275) | -14.34 (NA) — 1 participant analyzed
  Percent Change at Month 5: number analyzed (Participants) | 0 | 3 | 0
  Percent Change at Month 5 |  | -35.81 (9.326) |
  Percent Change at Month 6: number analyzed (Participants) | 0 | 2 | 0
  Percent Change at Month 6 |  | -33.56 (11.357) |

19. Secondary Outcome: Change From Baseline Over Time in Daily Rescue Analgesic Use Across Both Classes of Rescue Analgesics
Description: Based on average pill counts and assessed using a daily e-Diary. Permitted non-steroidal anti-inflammatory drugs (NSAIDs) included naproxen, ibuprofen, diclofenac, and celecoxib. Permitted opioids included hydrocodone + acetaminophen and codeine phosphate + acetaminophen.
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: pills/day
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
pills/day
  NSAID: Change at Month 1 | -0.84 (0.796) | 0.09 (0.388) | -0.67 (NA) — 1 participant analyzed
  NSAID: Change at Month 2: number analyzed (Participants) | 5 | 3 | 1
  NSAID: Change at Month 2 | -1.15 (0.785) | -0.17 (0.834) | 0.63 (NA) — 1 participant analyzed
  NSAID: Change at Month 3: number analyzed (Participants) | 2 | 3 | 1
  NSAID: Change at Month 3 | -0.96 (1.030) | -0.43 (1.091) | -0.71 (NA) — 1 participant analyzed
  NSAID: Change at Month 4: number analyzed (Participants) | 1 | 3 | 1
  NSAID: Change at Month 4 | -1.69 (NA) — 1 participant analyzed | 0.01 (0.845) | -0.63 (NA) — 1 participant analyzed
  NSAID: Change at Month 5: number analyzed (Participants) | 0 | 3 | 0
  NSAID: Change at Month 5 |  | 0.23 (1.197) |
  NSAID: Change at Month 6: number analyzed (Participants) | 0 | 2 | 0
  NSAID: Change at Month 6 |  | 0.63 (0.606) |
  Opioid: Change at Month 1 | 0.12 (0.552) | -0.06 (0.099) | -0.43 (NA) — 1 participant analyzed
  Opioid: Change at Month 2: number analyzed (Participants) | 5 | 3 | 1
  Opioid: Change at Month 2 | -0.17 (0.263) | -0.03 (0.049) | -0.51 (NA) — 1 participant analyzed
  Opioid: Change at Month 3: number analyzed (Participants) | 2 | 3 | 1
  Opioid: Change at Month 3 | -0.17 (0.242) | 0.02 (0.016) | -0.49 (NA) — 1 participant analyzed
  Opioid: Change at Month 4: number analyzed (Participants) | 1 | 3 | 1
  Opioid: Change at Month 4 | -0.34 (NA) — 1 participant analyzed | -0.01 (0.044) | -0.40 (NA) — 1 participant analyzed
  Opioid: Change at Month 5: number analyzed (Participants) | 0 | 3 | 0
  Opioid: Change at Month 5 |  | -0.05 (0.082) |
  Opioid: Change at Month 6: number analyzed (Participants) | 0 | 2 | 0
  Opioid: Change at Month 6 |  | 0.09 (0.121) |
  NSAID + Opioid: Change at Month 1 | -0.72 (1.178) | 0.03 (0.436) | -1.10 (NA) — 1 participant analyzed
  NSAID + Opioid: Change at Month 2: number analyzed (Participants) | 5 | 3 | 1
  NSAID + Opioid: Change at Month 2 | -1.33 (0.767) | -0.20 (0.830) | -1.14 (NA) — 1 participant analyzed
  NSAID + Opioid: Change at Month 3: number analyzed (Participants) | 2 | 3 | 1
  NSAID + Opioid: Change at Month 3 | -1.13 (1.273) | -0.41 (1.107) | -1.20 (NA) — 1 participant analyzed
  NSAID + Opioid: Change at Month 4: number analyzed (Participants) | 1 | 3 | 1
  NSAID + Opioid: Change at Month 4 | -2.03 (NA) — 1 participant analyzed | -0.00 (0.863) | -1.03 (NA) — 1 participant analyzed
  NSAID + Opioid: Change at Month 5: number analyzed (Participants) | 0 | 3 | 0
  NSAID + Opioid: Change at Month 5 |  | 0.18 (1.217) |
  NSAID + Opioid: Change at Month 6: number analyzed (Participants) | 0 | 2 | 0
  NSAID + Opioid: Change at Month 6 |  | 0.71 (0.485) |

20. Secondary Outcome: Number of Analgesic Use Responders and Non-Responders Over Time
Description: Based only on reduction of rescue analgesics used. Responders were defined as:
  * participants with no analgesic use at screening and no analgesic use added
  * participants with NSAID only use at screening and NSAID dose stopped, decreased, or stable (<15% increase) and no opioid use added
  * participants with opioid only use at screening and opioid dose stopped, decreased, or stable (<15% increase), opioid dose stopped and NSAID substituted (any dose), opioid dose decreased and NSAID added (any dose)
  * participants with NSAID + opioid use at screening and any of the following: NSAID dose stopped + opioid analgesic use stopped, decreased, or stable (<15% increase); NSAID dose decreased + opioid analgesic use stopped, decreased, or stable (<15% increase); NSAID dose stable (< 15% increase) + opioid analgesic use stopped, decreased, or stable (<15% increase); NSAID dose increased by >15% + opioid analgesic use stopped; NSAID dose increased by >15% + opioid analgesic dose decreases.
Time Frame: Months 1, 2, 3, 4, 5, 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
Participants
  Month 1: Responder | 5 | 2 | 1
  Month 1: Non-Responder | 2 | 1 | 0
  Month 2: Responder | 4 | 2 | 1
  Month 2: Non-Responder | 1 | 1 | 0
  Month 3: Responder | 2 | 1 | 1
  Month 3: Non-Responder | 0 | 2 | 0
  Month 4: Responder | 1 | 2 | 1
  Month 4: Non-Responder | 0 | 1 | 0
  Month 5: Responder | 0 | 2 | 0
  Month 5: Non-Responder | 0 | 1 | 0
  Month 6: Responder | 0 | 0 | 0
  Month 6: Non-Responder | 0 | 2 | 0

21. Secondary Outcome: Patient Global Impression of Change (PGIC) Scores Over Time
Description: The PGIC is a 7-point response scale where participants rate their endometriosis related pain as: very much improved (1), much improved (2), minimally improved (3), not changed (4), minimally worse (5), much worse (6), very much worse (7).
Time Frame: Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Month 1 | 2.9 (1.35) | 2.3 (0.58) | 2.0 (NA) — 1 participant analyzed
  Month 2: number analyzed (Participants) | 2 | 3 | 1
  Month 2 | 2.0 (0.00) | 1.3 (0.58) | 2.0 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 1 | 3 | 1
  Month 3 | 2.0 (NA) — 1 participant analyzed | 2.0 (1.00) | 5.0 (NA) — 1 participant analyzed
  Month 4: number analyzed (Participants) | 0 | 3 | 1
  Month 4 |  | 2.0 (1.00) | 2.0 (NA) — 1 participant analyzed
  Month 5: number analyzed (Participants) | 0 | 2 | 0
  Month 5 |  | 2.5 (0.71) |
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 1.0 (NA) — 1 participant analyzed |

22. Secondary Outcome: Overall Endometriosis-Associated Pain Via NRS (7-Day Recall) Scores Over Time
Description: The endometriosis-associated pain questionnaire is an 11-point NRS assessing overall endometriosis-associated pain over a 7-day recall period. Participants assessed their endometriosis-associated pain on a scale of 0 to 10, with 0 = no pain and 10 = worst pain ever.
Time Frame: Month 0 (baseline), Months 1, 2, 3, 4, 5, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline: number analyzed (Participants) | 5 | 3 | 1
  Baseline | 8.2 (1.79) | 9.0 (1.00) | 7.0 (NA) — 1 participant analyzed
  Month 1 | 5.7 (3.04) | 7.7 (1.15) | 8.0 (NA) — 1 participant analyzed
  Month 2: number analyzed (Participants) | 2 | 3 | 1
  Month 2 | 4.5 (0.71) | 2.7 (1.15) | 5.0 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 1 | 3 | 1
  Month 3 | 9.0 (NA) — 1 participant analyzed | 5.3 (2.31) | 8.0 (NA) — 1 participant analyzed
  Month 4: number analyzed (Participants) | 0 | 3 | 1
  Month 4 |  | 3.3 (0.58) | 7.0 (NA) — 1 participant analyzed
  Month 5: number analyzed (Participants) | 0 | 2 | 0
  Month 5 |  | 8.0 (0.00) |
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 4.0 (NA) — 1 participant analyzed |

23. Secondary Outcome: Endometriosis Health Profile-30 (EHP-30) Scores Over Time: Pain
Description: The EHP-30 is a disease-specific self-administered questionnaire used to measure health-related quality of life in women with endometriosis. Domains used in the study included Pain, Control and Powerlessness, Well-Being, Social Support, Self-Image, and Sexual Intercourse. Each domain is calculated on a scale from 0 = best possible health status to 100 = worst possible health status.
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 59.42 (11.694) | 47.73 (14.193) | 59.09 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 38.07 (26.529) | 17.42 (22.422) | 38.64 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 27.27 (NA) — 1 participant analyzed |

24. Secondary Outcome: EHP-30 Scores Over Time: Control and Powerlessness
Description: as for outcome 23
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 71.43 (19.159) | 56.94 (19.691) | 41.67 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 36.46 (32.874) | 26.39 (21.382) | 25.00 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 8.33 (NA) — 1 participant analyzed |

25. Secondary Outcome: EHP-30 Scores Over Time: Emotional Well-Being
Description: as for outcome 23
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 29.76 (8.815) | 50.00 (8.333) | 45.83 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 18.75 (12.500) | 23.61 (17.347) | 37.50 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 25.00 (NA) — 1 participant analyzed |

26. Secondary Outcome: EHP-30 Scores Over Time: Social Support
Description: as for outcome 23
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 48.21 (21.565) | 45.83 (19.094) | 50.00 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 17.19 (11.831) | 16.67 (28.868) | 18.75 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 25.00 (NA) — 1 participant analyzed |

27. Secondary Outcome: EHP-30 Scores Over Time: Self-Image
Description: as for outcome 23
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 50.00 (22.048) | 36.11 (31.549) | 75.00 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 43.75 (41.597) | 8.33 (14.434) | 8.33 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 3 | 0
  Month 6 |  | 16.67 (NA) — 1 participant analyzed |

28. Secondary Outcome: EHP-30 Scores Over Time: Sexual Intercourse
Description: as for outcome 23
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6 | 2 | 1
score on a scale
  Baseline | 70.00 (22.361) | 62.50 (31.820) | 60.00 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 2 | 1
  Month 3 | 45.00 (23.452) | 45.00 (42.426) | 60.00 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 30.00 (NA) — 1 participant analyzed |

29. Secondary Outcome: EuroQol-5D 5 Level (EQ-5D-5L) Scores Over Time: Mobility
Description: The EQ-5D-5L is a health state utility instrument with 5 items that comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each of which is rated on 5 levels of severity (1=no problem, 2=slight problems, 3=moderate problems, 4=severe problems, 5=extreme problems) and a separate visual analog scale (VAS) indicating a participant's rating of their current health status (health today) on a scale of from 0 (worst health imaginable) to 100 (best health imaginable).
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 1.4 (0.53) | 1.0 (0.00) | 1.0 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 1.3 (0.50) | 1.0 (0.00) | 2.0 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 1.0 (NA) — 1 participant analyzed |

30. Secondary Outcome: EQ-5D-5L Scores Over Time: Self-Care
Description: as for outcome 29
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 1.0 (0.00) | 1.0 (0.00) | 1.0 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 1.0 (0.00) | 1.0 (0.00) | 1.0 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 1.0 (NA) — 1 participant analyzed |

31. Secondary Outcome: EQ-5D-5L Scores Over Time: Usual Activities
Description: as for outcome 29
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 2.0 (0.82) | 1.3 (0.58) | 1.0 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 1.5 (0.58) | 1.7 (1.15) | 2.0 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 1.0 (NA) — 1 participant analyzed |

32. Secondary Outcome: EQ-5D-5L Scores Over Time: Pain/Discomfort
Description: as for outcome 29
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 2.7 (0.76) | 2.7 (0.58) | 4.0 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 2.0 (1.15) | 1.7 (0.58) | 3.0 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 1.0 (NA) — 1 participant analyzed |

33. Secondary Outcome: EQ-5D-5L Scores Over Time: Anxiety/Depression
Description: as for outcome 29
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 1.0 (0.00) | 1.3 (0.58) | 1.0 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 1.0 (0.00) | 1.0 (0.00) | 1.0 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 1.0 (NA) — 1 participant analyzed |

34. Secondary Outcome: EQ-5D-5L VAS Scores Over Time: Health Today
Description: The EQ-5D-5L is a health state utility instrument with 5 items that comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each of which is rated on 5 levels of severity (1=no problem, 2=slight problems, 3=moderate problems, 4=severe problems, 5=extreme problems) and a separate VAS indicating a participant's rating of their current health status (health today) on a scale of from 0 (worst health imaginable) to 100 (best health imaginable).
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 79.7 (15.16) | 53.3 (35.12) | 72.0 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 72.8 (17.63) | 85.0 (15.00) | 70.0 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 94.0 (NA) — 1 participant analyzed |

35. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) Scores Over Time: Percent Work Missed Due to Problem
Description: Absenteeism is presented as the mean percentage of work time missed due to health problem (as reported on the WPAI:SHP), and is calculated as: 100*number of hours of work missed due to health problem / (number of hours of work missed due to health problem + number of hours worked). WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Month 0 (baseline), Month 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percent of work time missed
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6 | 3 | 0
percent of work time missed
  Baseline | 0.16 (0.205) | 0.08 (0.144) |
  Month 6: number analyzed (Participants) | 3 | 1 | 0
  Month 6 | 0.00 (0.000) | 0.00 (NA) — 1 participant analyzed |

36. Secondary Outcome: WPAI:SHP Scores Over Time: Percent Impairment While Working Due to Problem
Description: Presenteeism (the extent to which health problem decreased productivity) is presented as the mean percentage of impairment while working due to health problem, and is calculated as: 100*scale value of question 5 on the WPAI (between 0 and 10) / 10. WPAI:SHP is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Month 0 (baseline), Month 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percent impairment while working
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6 | 3 | 0
percent impairment while working
  Baseline | 0.57 (0.273) | 0.53 (0.153) |
  Month 6: number analyzed (Participants) | 3 | 1 | 0
  Month 6 | 0.30 (0.265) | 0.30 (NA) — 1 participant analyzed |

37. Secondary Outcome: WPAI:SHP Scores Over Time: Percent Overall Work Impairment Due to Problem
Description: The mean percentage of overall work impairment due to health problem (based on the WPAI questionnaire) is presented, and is calculated as: Absenteeism (%) + extent to which health problem decreased productivity (%)* [number of hours worked / (number of hours of work missed due to health problem + number of hours worked)]. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Month 0 (baseline), Month 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percent overall work impairment
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6 | 3 | 0
percent overall work impairment
  Baseline | 0.61 (0.307) | 0.56 (0.194) |
  Month 6: number analyzed (Participants) | 3 | 1 | 0
  Month 6 | 0.30 (0.265) | 0.30 (NA) — 1 participant analyzed |

38. Secondary Outcome: WPAI:SHP Scores Over Time: Percent Activity Impairment Due to Problem
Description: Activity impairment due to health problem (the extent to which health problem affected the ability to perform usual daily activities) is presented as the mean percentage of activity impairment, and is calculated as 100*scale value of WPAI question 6 (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Month 0 (baseline), Month 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage impairment of activity
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
percentage impairment of activity
  Baseline | 0.66 (0.237) | 0.67 (0.058) | 0.70 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 3 | 1 | 1
  Month 6 | 0.40 (0.346) | 0.30 (NA) — 1 participant analyzed | 0.70 (NA) — 1 participant analyzed

39. Secondary Outcome: Health Endometriosis Treatment Satisfaction Questionnaire (ETSQ) Scores Over Time
Description: The 6-item ETSQ was developed to assess patient-reported satisfaction with effects on endometriosis pain, dysmenorrhea, dyspareunia, amount of bleeding tolerability and overall treatment satisfaction. The ETSQ has a 7 point response scale. The range for this scale is 0 to 36, with lower ETSQ scores reflecting lower levels of satisfaction with endometriosis treatment.
Time Frame: Month 0 (baseline), Months 3, 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 19.71 (4.536) | 18.00 (0.000) | 18.00 (NA) — 1 participant analyzed
  Month 3: number analyzed (Participants) | 4 | 3 | 1
  Month 3 | 22.25 (9.430) | 25.47 (6.652) | 25.00 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 0 | 1 | 0
  Month 6 |  | 31.00 (NA) — 1 participant analyzed |

40. Secondary Outcome: PROMIS Fatigue Short Form 6a Scores Over Time
Description: The PROMIS Fatigue Short Form 6a is self-administered and composed of 6 questions to evaluate fatigue. Possible scores range from 6 to 30, 6 = not at all (no fatigue), and 30 = very much (most fatigue).
Time Frame: Month 0 (baseline), Month 6
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 3 | 1
score on a scale
  Baseline | 22.1 (4.10) | 19.3 (6.11) | 27.0 (NA) — 1 participant analyzed
  Month 6: number analyzed (Participants) | 3 | 1 | 1
  Month 6 | 15.3 (7.77) | 11.0 (NA) — 1 participant analyzed | 21.0 (NA) — 1 participant analyzed

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 6 months, plus 30 days.
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/7 | 3/3 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=7) | Group B (N=3) | Group C (N=1)
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
GARDNERELLA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VAGINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
POLYDIPSIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
IRRITABILITY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ADNEXA UTERI PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
MENSTRUATION DELAYED (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to early study termination at Treatment Month 6 with low subject enrollment, no clinically or statistically meaningful efficacy conclusions can be made. The study was terminated early for business reasons, not for safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT03343067/Prot_SAP_000.pdf